CLINICAL TRIAL: NCT03492034
Title: Insertion of Intrauterine Contraceptive Device During Cesarean Section: Randomized Clinical Trial
Brief Title: IUD Insertion During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AS1750
Record Dates: First submitted 2018-03-24; First posted 2018-04-10 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IUD during CS (Active Comparator)
  Interventions: Device: IUD during CS
- IUD after puerperium (Active Comparator)
  Interventions: Device: IUD after puerperium

INTERVENTIONS:
Device: IUD during CS — IUD insertion during CS
  Arms: IUD during CS
Device: IUD after puerperium — IUD after puerperium
  Arms: IUD after puerperium

SUMMARY:
Insertion of Intrauterine Contraceptive Device during Cesarean Section: Randomized Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant woman aged between 18 to 40 years old.
2. Scheduled for elective cesarean section at gestational age between 37 to 42 weeks.
3. Body mass index between 19-30 kg/m2
4. Seeking contraception after delivery.

Exclusion Criteria:

1. History of menorrhagia or severe dysmenorrhea.
2. History of pelvic inflammatory disease or current pelvic infection (ex: puerperal sepsis, purulent cervicitis).
3. Patients who have bleeding disorders.
4. Anemia (Hb < 9 g %).
5. Chronic depilating diseases reducing immunity such as Diabetes.
6. Structural uterine anomaly or large uterine fibroids distorting anatomy.
7. History of previous IUD expulsion or removal for complications.
8. Unexplained uterine bleeding.
9. Copper allergy or Wilson disease.
10. Gestational trophoblastic disease with persistently elevated Beta HCG.
11. Predisposing factor to postoperative infection (e.g. rupture of membranes prior to admission or delivery of a stillborn baby at cesarean section).
12. Complications during cesarean section e.g. postpartum hemorrhage.
13. Cesarean section during placenta previa.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
IUD expulsion rate | 6 weeks

SECONDARY OUTCOMES:
Bleeding | 6 weeks
  number of pads changed per day
Degree of Pain | 6 weeks
  Visual Analogue Scale from 1 to10 (0 being no pain and 10 maximum pain tolerated)
dyspareunia | 6 weeks
  Visual Analogue Scale from 0 to10 (0 being no pain and 10 maximum pain tolerated)
patient satisfaction | 6 weeks
  Visual Analogue Scale from 0 to10 (0 being maximum dis-satisfaction and 10 maximum satisfaction)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

REFERENCES:
- [Derived] Sothornwit J, Kaewrudee S, Lumbiganon P, Pattanittum P, Averbach SH. Immediate versus delayed postpartum insertion of contraceptive implant and IUD for contraception. Cochrane Database Syst Rev. 2022 Oct 27;10(10):CD011913. doi: 10.1002/14651858.CD011913.pub3. PMID 36302159